CLINICAL TRIAL: NCT00340626
Title: Genetic Analysis of Hereditary Non-Syndromic Oral Clefts
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999997035; OH97-HG-N035
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Hereditary Oral Clefts
Keywords: Linkage Analysis; Genotyping; Birth Defects; Family Study; Positional Cloning
MeSH Terms: conditions — Congenital Abnormalities

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, saliva

GROUPS / COHORTS (2):
- Control: healthy individuals with no history of oral cleftsto serve as controls
- Oral Cleft Family Members: individuals with unilateral or bilateral cleft lip with or without cleft palate and their unaffected relatives

SUMMARY:
In a collaborative effort with the IBN AL-NAFEES Hospital (Damascus, Syrian Arab Republic), individuals from multiplex families determined to have hereditary oral clefts will be studied. The purpose of this study is to identify the gene(s) involved in heritable oral clefts by linkage analysis and gene mapping strategies. Characterization of genes involved in inherited oral clefts could provide important insight into the inheritance and pathogenesis of this disease.

DETAILED DESCRIPTION:
In a collaborative effort with the IBN AL-NAFEES Hospital (Damascus, Syrian Arab Republic), individuals from multiplex families determined to have hereditary oral clefts will be studied. Healthy Syrian individuals with no family history of oral clefts will also be enrolled as a comparison group. The purpose of this study is to identify the gene(s) involved in heritable oral clefts by linkage analysis and gene mapping strategies. Characterization of genes involved in inherited oral clefts could provide important insight into the inheritance and pathogenesis of this disease. All families are enrolled into the study by our Syrian collaborators (under Ethics Board approval from the IBN AL-NAFEES Hospital) and only coded phenotype data and coded biospecimens are ever received at the NIH.

ELIGIBILITY:
* INCLUSION CRITERIA:

Enrollment in this study will be limited to individuals with non-syndromic unilateral or bilateral cleft lip with or without cleft palate and their unaffected relatives, from families which meet the following criteria:

1. A cluster of 2 or more affected first degree relatives, such as a parent and two offspring or 2 siblings, or
2. The occurrence of oral clefts in each of 2 generations in either the proband's paternal or maternal lineages.
3. The occurrence of oral clefts in 2 or more cousins (up to second cousins)

The subject population is comprised of probands and their families previously examined at the IBN-AL NAFEES Hospital or at other hospitals and clinics in the Syrian Arab Republic as well

as healthy controls from the same population. Consent documents are in Arabic language for non-English-speaking subjects

EXCLUSION CRITERIA:

Individuals unable to provide consent, except for cases who are children and mentally impaired persons with consenting parents or guardians.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: individuals with unilateral or bilateral cleft lip with or without cleft palate and their unaffected relatives@@@
Sampling Method: Non-Probability Sample
Enrollment: 690 (Actual)
Dates: Start 1997-08-31 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-03-12 (Actual)

PRIMARY OUTCOMES:
Identification of genetic risk variants for oral clefts | Ongoing
  To identify and characterize genes responsible for non- syndromic and syndromic oral clefts by genetic family studies including linkage analysis, association analysis, positional cloning, evaluation of candidate genes, and eventual evaluation of mutations in identified genes.

CONTACTS AND LOCATIONS:
Overall Officials: Joan Bailey-Wilson, Ph.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- IBN Al Nafees Hospital, Damascus, Syria

REFERENCES:
- [Background] Wyszynski DF, Beaty TH, Maestri NE. Genetics of nonsyndromic oral clefts revisited. Cleft Palate Craniofac J. 1996 Sep;33(5):406-17. doi: 10.1597/1545-1569_1996_033_0406_gonocr_2.3.co_2. PMID 8891372
- [Background] Zlotogora J. Genetic disorders among Palestinian Arabs: 1. Effects of consanguinity. Am J Med Genet. 1997 Feb 11;68(4):472-5. doi: 10.1002/(sici)1096-8628(19970211)68:43.0.co;2-o. PMID 9021024
- [Background] Shprintzen RJ, Siegel-Sadewitz VL, Amato J, Goldberg RB. Anomalies associated with cleft lip, cleft palate, or both. Am J Med Genet. 1985 Apr;20(4):585-95. doi: 10.1002/ajmg.1320200404. PMID 3993684